CLINICAL TRIAL: NCT06768866
Title: Factors Influencing Postsurgical Acute Pain and Its Pharmacological Management Among Patient Undergoing Elective Surgeries at Tertiary Care Hospital Mardan
Brief Title: Factors Influencing PAP and Its PM Among Patient Undergoing Elective Surgeries at Tertiary Care Hospital Mardan
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/025
Record Dates: First submitted 2024-12-18; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Surgery-Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Gruop 1 — To determine factors influencing Postsurgical acute pain

SUMMARY:
Postsurgical acute pain is a critical factor impacting recovery, patient satisfaction, and the risk of complications in surgical patients. Effective pain management is essential for enhancing patient outcomes and reducing the likelihood of chronic pain development.

DETAILED DESCRIPTION:
However, pain perception is influenced by various factors, including demographic characteristics, types, duration and complexity of surgery, and pharmacological approaches. This study aims to identify these contributing factors and assess the effectiveness of different analgesics in managing postsurgical pain in a tertiary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ages of 18 years and above.
* ASA Class I,II are scheduled for elective surgeries under general anesthesia at Tertiary care hospital Mardan.

Exclusion Criteria:

* Chronic opioid and NSAID user, tricyclic antidepressants and selective serotonin reuptake inhibitors.
* People with bleeding disorders.
* Postoperative respiratory depression, patient with emergency surgeries or admitted to ICU Postoperative.
* Procedure perform under regional Anesthesia, history of hypersensitivity to analgesic drugs and refusal to participate"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To determine factors influencing Postsurgical acute pain
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 12 Months
  Visual analog scale (0-10 VAS)and it was categorized using the following terms : no pain (0), mild (1-3), moderate (4-6),severe (7-9),or worse pain (10)

CONTACTS AND LOCATIONS:
Locations (1):
- Mardan Medical Complex, Mardan, Khyber Pakhtunkhwa, Pakistan